CLINICAL TRIAL: NCT01836601
Title: The Effect of a Family-Centered Nighttime Communication Bundle on Shared Mental-Model Building, Safety, and Patient Experience
Brief Title: Nighttime Communication Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Program for Patient Safety and Quality (Unknown)
Responsible Party: Principal Investigator, Alisa Khan, Instructor, Pediatrics, Boston Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-P00006501
Record Dates: First submitted 2013-04-10; First posted 2013-04-22 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Communication
Keywords: safety; patient experience; family-centered rounds
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-nighttime communication intervention arm (No Intervention): This arm is the pre-intervention arm of parents, nurses, and residents before the nighttime communication bundle has been enacted.
- Post-nighttime communication intervention arm (Experimental): This arm is the post-intervention arm of parents, nurses, and residents after the nighttime communication bundle has been enacted.
  Interventions: Behavioral: Family-centered nighttime communication bundle

INTERVENTIONS:
Behavioral: Family-centered nighttime communication bundle
  Arms: Post-nighttime communication intervention arm

SUMMARY:
This study seeks to determine whether a family-centered nighttime communication intervention improves: 1) shared understanding by parents, residents, and nurses of hospitalized pediatric patient's medical plans, 2) parent-reported errors, 3) parent and provider experience of nighttime medical care.

ELIGIBILITY:
Inclusion Criteria:

* Parents of patients admitted to the general pediatrics inpatient units
* Overnight nurses working on the general pediatrics inpatient units
* Overnight residents working on the general pediatrics inpatient units

Exclusion Criteria:

* Non-English speaking parents

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1334 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Concordance between parent, resident, and nurse reported elements of the patient action plan and overall plan | 18 months
  This will be assessed through surveys administered to parents, residents, and nurses for a subset of patients every evening. Parent, resident, and nurse responses will be compared pre and post-intervention.

SECONDARY OUTCOMES:
Parent-reported medical errors | 18 months
  This will be assessed through surveys administered to parents for a subset of patients every evening. Parent error reporting will be compared pre and post-intervention.

OTHER OUTCOMES:
Provider and parent experience of nighttime care | 18 months
  This will be assessed through surveys administered to parents and providers for a subset of patients. Answers will be compared pre and post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Khan A, Rogers JE, Forster CS, Furtak SL, Schuster MA, Landrigan CP. Communication and Shared Understanding Between Parents and Resident-Physicians at Night. Hosp Pediatr. 2016 Jun;6(6):319-29. doi: 10.1542/hpeds.2015-0224. PMID 27188189